CLINICAL TRIAL: NCT02830789
Title: Investigation of the Optimal Calcium Supplement Following Roux-en-Y Gastric Bypass in Order to Treat Secondary Hyperparathyroidism: A Clinical Randomized Trial
Brief Title: Investigation of the Optimal Calcium Supplement Following Roux-en-Y Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Lene Ring Madsen, PhD student, MD, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20160610
Record Dates: First submitted 2016-07-06; First posted 2016-07-13 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Roux-en-Y Gastric Bypass; Hyperparathyroidism, Secondary
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — Calcium Carbonate; Calcium Citrate; Gastric Bypass

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcium Carbonate (Experimental): 1 tablet Unikalk Forte + 1 placebo tablet by mouth three times daily equal to 1200 mg elementary calcium and 57 µg Vitamin D3
  Interventions: Dietary Supplement: Calcium Carbonate; Dietary Supplement: Placebo; Procedure: Roux-en-Y gastric bypass
- Calcium Citrate (Experimental): 2 tablets Unikalk Citrat by mouth three times daily equal to 1200 mg elementary calcium and 60 µg Vitamin D3
  Interventions: Dietary Supplement: Calcium Citrate; Procedure: Roux-en-Y gastric bypass

INTERVENTIONS:
Dietary Supplement: Calcium Carbonate
  Other Names: Unikalk Forte
  Arms: Calcium Carbonate
Dietary Supplement: Calcium Citrate
  Other Names: Unikalk Citrat
  Arms: Calcium Citrate
Dietary Supplement: Placebo — Tablet manufactured to mimic a calcium carbonate tablet
  Arms: Calcium Carbonate
Procedure: Roux-en-Y gastric bypass — Roux-en-Y gastric bypass surgery at least 12 months before study inclusion

SUMMARY:
This study investigates whether calcium citrate or calcium carbonate are the optimal supplement to treat secondary hyperparathyroidism following Roux-en-Y gastric bypass operation.

Half of the participants will be randomized to receive calcium citrate, while the other half will receive calcium carbonate. The study will be double blinded.

ELIGIBILITY:
Inclusion Criteria:

* Roux-en-Y gastric bypass operation ≥12 months ago
* Parathyroid hormone > 6.9 pmol/l
* Vitamin D > 50 nmol/l
* P-Calcium [1.18-1.32] mmol/l

Exclusion Criteria:

* Liver disease
* Renal disease
* Hypercalcemia
* Untreated thyroid disease
* Parathyroid disease except secondary hyperparathyroidism
* Use of diuretics, bisphosphonates, calcitonin, teriparatide, oral corticosteroids, anabolic steroids, calcimimetics, lithium, strontium, denosumab or anticonvulsants within 1 year of inclusion
* abusing alcohol

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-12; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Parathyroid Hormone | Change from baseline at 6 weeks and 12 weeks

SECONDARY OUTCOMES:
Se-ion-calcium | Change from baseline at 6 weeks and 12 weeks
P-magnesium | Change from baseline at 6 weeks and 12 weeks
P-phosphate | Change from baseline at 6 weeks and 12 weeks
P-25-OH-vitamin D | Change from baseline at 6 weeks and 12 weeks
P-calcitriol | Change from baseline at 6 weeks and 12 weeks
P-24,25-(OH)2-vitamin D | Change from baseline at 6 weeks and 12 weeks
Vitamin D binding protein | Change from baseline at 6 weeks and 12 weeks
Procollagen type 1 N-terminal propeptide (P1NP) | Change from baseline at 6 weeks and 12 weeks
P-bone specific alkaline phosphatase | Change from baseline at 6 weeks and 12 weeks
Cross-linked C-telopeptide (CTX) | Change from baseline at 6 weeks and 12 weeks
24h U-calcium | Change from baseline at 12 weeks
24h U-phosphate | Change from baseline at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Enodocrinology and Internal Medicine, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No